CLINICAL TRIAL: NCT05758038
Title: US-guided Radiofrequency Ablation Versus Microwave Ablation in the Treatment of Benign Thyroid Nodules
Brief Title: US-guided RFA vs MWA in the Treatment of Benign Thyroid Nodules
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Gamal Mokhtar, Assistant Lecturer, Assiut University
Other Study IDs: RFA/MWA in thyroid nodules.
Record Dates: First submitted 2023-02-12; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Thyroid Nodule (Benign)
MeSH Terms: conditions — Thyroid Nodule | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: Patients with benign thyroid nodules undergo RFA
  Interventions: Procedure: Radiofrequency ablation/Microwave ablation
- group 2: Patients with benign thyroid nodule undergo MWA
  Interventions: Procedure: Radiofrequency ablation/Microwave ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation/Microwave ablation — thermal ablation by radiofrequency and Microwave

SUMMARY:
To evaluate the clinical outcomes of RFA and MWA for benign thyroid nodules treatment

DETAILED DESCRIPTION:
The thyroid nodule is one of the most common lesions in clinical practice and has been increasingly detected in approximately 50% of the general population by ultrasound (US) examination in the past two decades due to the widespread use of radiological imaging.

Benign thyroid nodules (BTNs) proven cytologically by fine-needle aspiration biopsy (FNAB) account for 85 to 95% of all thyroid nodules.

Despite the fact that the majority of thyroid nodules diagnosed are benign and do not cause significant clinical symptoms, some nodules may lead to compression-related symptoms. In addition, thyrotoxic symptoms may develop due to hyperfunctioning of some nodules.

To date, surgical resection is the main treatment for thyroid nodules. However, it has serious drawbacks such as leading to excessive surgical trauma or hypothyroidism, influencing the aesthetic aspect of the neck, or increasing a post-operative recurrence rate.

RFA has shown good efficacy and safety in the management of thyroid nodule related cosmetic problems and pressure symptoms.

MWA is a newly developed local thermal ablation technique that has fast heating speed, strong coagulation ability and large ablation zone, and has become a great therapeutic method in heat ablation therapy (8) The advantages of ultrasound-guided minimally invasive ablation therapy over the traditional surgery include simpler operation and shorter treatment time. (8)

ELIGIBILITY:
Inclusion Criteria:

* Solid or mixed nodules with predominant solid component with benign pathological result from US guided fine needle aspiration (FNAC).
* Symptomatic and/or cosmetic problems.
* Clinical thyrotoxicosis and hyperthyroidism caused by autonomously functioning thyroid nodules (AFTNs)
* Refusal or ineligible for surgery.
* Anxiety about a malignant transformation.

Exclusion Criteria:

* Malignant nodules on US.
* Cytological evidence for malignancy
* Patients with abnormal coagulation profile.
* previous surgery or medicine for the thyroid, and vocal cord palsy in the side contralateral to the target nodules.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with benign thyroid nodules come to assiut university hospital for treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
symptoms score | 2 years
  symptoms score will be assessed by (visual analogue scale) a score from 1 to 10 will be given by the patient according to each symptom including (neck pain , dysphagia , foreign body sensation , discomfort and cough)
  1 is the minimum score indicating the best outcome and 10 is the maximum score indicating worst outcome
thyroid nodule volume reduction | 2 years
  volume reduction ratio VRR assessed by Ultrasound = [(initial volume - final volume)/initial volume] x 100.
cosmetic score | 2 years
  cosmetic score will be measured by the physician (1, no palpable mass; 2, no cosmetic problem but palpable mass; 3, a cosmetic problem on swallowing only; and 4, a readily detected cosmetic problem)
  1 indicates the best outcome and 4 indicates the worst outcome

CONTACTS AND LOCATIONS:
Overall Officials: Omar Mokhtar, Assistant lecturer, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Russ G, Ben Hamou A, Poiree S, Ghander C, Menegaux F, Leenhardt L, Buffet C. Learning curve for radiofrequency ablation of benign thyroid nodules. Int J Hyperthermia. 2021;38(1):55-64. doi: 10.1080/02656736.2021.1871974. PMID 33491515
- [Background] Liu YJ, Qian LX, Liu D, Zhao JF. Ultrasound-guided microwave ablation in the treatment of benign thyroid nodules in 435 patients. Exp Biol Med (Maywood). 2017 Sep;242(15):1515-1523. doi: 10.1177/1535370217727477. Epub 2017 Aug 28. PMID 28847173
- [Background] Erturk MS, Cekic B, Celik M. Microwave Ablation of Benign Thyroid Nodules: Effects on Systemic Inflammatory Response. J Coll Physicians Surg Pak. 2020 Jul;30(7):694-700. doi: 10.29271/jcpsp.2020.07.694. PMID 32811597
- [Background] Deandrea M, Trimboli P, Garino F, Mormile A, Magliona G, Ramunni MJ, Giovanella L, Limone PP. Long-Term Efficacy of a Single Session of RFA for Benign Thyroid Nodules: A Longitudinal 5-Year Observational Study. J Clin Endocrinol Metab. 2019 Sep 1;104(9):3751-3756. doi: 10.1210/jc.2018-02808. PMID 30860579